CLINICAL TRIAL: NCT02666989
Title: Open-Label Placebo for the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Ziv Carmel, psychiatrists, Shalvata Mental Health Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Yehuda04
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Placebo; Open-label; Clinical practice
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- open placebo (Active Comparator): 8 weeks of open placebo treatment
  Interventions: Drug: placebo
- waitlist group (No Intervention): 4 weeks of waiting list followed by 4 weeks of open placebo treatment

INTERVENTIONS:
Drug: placebo — 2 placebo pills twice a day
  Arms: open placebo

SUMMARY:
Open label placebo treatment has been tried for irritable bowel syndrome (Kaptchuk et al, 2010), where three weeks of open label placebo proved superior to a wait-listed control group. Another pilot study demonstrated efficacy in treating children suffering from ADHD with open label placebo treatment (Sandler & Bodfish, 2007). Recent work has shown that placebo openly given can have significant analgesic effects for acute migraines (Kam-Hansen et al, 2014) and for experimentally-induced pain (Schafer at al, 2015). A preliminary attempt to treat depression with open label placebo proved the feasibility of such a study, but was too small and brief for conclusive results (Kelley et al, 2012).

We provide here the protocol for a study to assess the effect of open label placebo treatment for depression.

DETAILED DESCRIPTION:
participants will be recruited through advertisements in the traditional and on-line press, and via mental health care workers in local clinics. The psychiatrists in the study team will also have the option to access to the waiting list of outpatient clinics at the Shalvata Mental Health Center, and recruit patients (who's intake appointment in the outpatient clinic is expected to take place in more than 2 months) to the study via phone or face to face in the clinic. If a subject is already taking antidepressant treatment he can be recruited immediately to the study. If a subject is not taking an antidepressant treatment, and in his examination he is diagnosed with depression, the investigator will advice him to approach an outpatient clinic and start taking antidepressant medication. If the subjects refuses to use medications he will be recruited to the study medication-free.

Patients will be invited to participate in the study and the following wording will be used:

"we invite you to participate in a novel mind-body study harnessing placebo effects for the treatment of depression. In the study you will recieve, either immediately or following a waiting period, placebo (inert) tablets. There will be no active component in the tablet, but there is a good chance that it will alleviate some of the depressive symptoms. Furthermore, recent scientific evidence suggests that placebo tablets can initiate healthy responses even if a person knows they are placebos".

Each participant will provide signed informed consent. Each subject will receive a letter to his personal physician or psychiatrist in the community/hospital. Additionally, the study team will also contact the personal physician and inform him of the study. Subjects will continue their psychiatric follow-up and treatment as usual during the whole period of the study. If the study team recognized a suicidal deterioration the personal physician/psychiatrist will be notified immediately via phone. If a subject is currently without psychiatric follow-up, he will examined during the assessment points (every 2 weeks) of the study protocol by one of the physicians of the study team.

Before the first session, each participant will be randomized to one of two possible interventions: either 8 weeks of open label placebo, or 4 weeks of waitlist followed by four weeks of open label placebo.

The randomization procedure will be stratified to account for two groups of subjects: those currently on a stable dose of medication, and those currently receiving no medication. Therefore, each time a subject from one of these groups is randomized to one of the two interventions (open label placebo or wait list), the next subject from the same group will be assigned to the other intervention. By this method, we will obtain the same proportion of medicated and unmedicated patients in each of the two intervention arms.

At the first session, the participant positive expectation and commitment will be promoted by discussing with the participant the following four points: (a) in research, placebos have been found to be safe in terms of side-effects and roughly 80% as effective as antidepressants; (b) recent research suggests that a patient can benefit from a placebo even when he knows that he is taking a placebo; (c) placebos appear to promote automatic self-healing processes, possibly through classical conditioning ; just taking tablets can cause the release of neurotransmitters and activate specific regions of the brain related to depression] (d) placebo-treated patients who adhere to the tablet regimen have better outcomes, and therefore the placebos should be taken faithfully, and (e) positive expectations enhance placebo effects, but it is perfectly normal to have doubts or disbelief and won't interfere with the effect.

At the end of the first session, the researcher will open an envelope which will reveal to researcher and participant to which group the latter has been randomized. Both treatment arm and no-treatment control will have identical patient-provider interactions and be of equal length. Those in the waitlist group will be encouraged to continue in the study.

The placebo will be a colored tablet. Each participant will be enjoined to take two capsules in the morning, and two in the evening.

After four weeks, the placebo group will continue with a second four week period of placebo treatment, and the waitlist group will start to receive 4 weeks of placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

i. Major Depressive Episode according to DSM-V ii. Mild to Moderate depression (8>HAM-D-17 <24) iii. Receiving antidepressant medication with no change in medication in the last two weeks or not receiving antidepressants medication

Exclusion Criteria:

i. Psychotic depression ii. Agitated depression iii. Bipolar depression iv. Current suicidality or past suicide attempt v. Current drug or alcohol abuse vi. Psychotic disorder vii. Drug and/or alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
v. HAM-D-17 (Hamilton, 1960) | 8 weeks